CLINICAL TRIAL: NCT02415621
Title: A Pilot Study of Adaptive Abiraterone Therapy for Metastatic Castration Resistant Prostate Cancer
Brief Title: Adaptive Abiraterone Therapy for Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17981
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: metastatic; castration resistant; abiraterone therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone Acetate Therapy (Other): Study schedule involves stopping FDA Approved abiraterone after participants achieve a good PSA response (50% or more decline of pre-abiraterone PSA) and then restarting abiraterone after their PSA reaches the level of pre-abiraterone PSA.
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — 1000 mg by mouth (PO) every day (QD)
  Other Names: Zytiga

SUMMARY:
Abiraterone is approved in the United States by the U.S. Food and Drug Administration (FDA) to treat metastatic prostate cancer at 1000 mg daily.

The purpose of this study is to find out if an on and off schedule of taking abiraterone would prolong the participant's cancer's response to this drug and maintain their functionality to perform their daily activities.

DETAILED DESCRIPTION:
In this pilot study, 10 black participants and 15 non-black participants will be enrolled after achieving 50% or more decline of their prostatic specific antigen (PSA) while on abiraterone for asymptomatic or minimally symptomatic metastatic castration resistant prostate cancer (mCRPC). Abiraterone will be stopped and will not be re-initiated until there is 50% or more increase of the PSA. Each time abiraterone is stopped, it will be defined as the start of a new adaptive therapy cycle. Participants who cannot achieve a 50% decline of their PSA after restarting abiraterone will continue abiraterone until they develop radiographic disease progression. If the decline in performance status does not occur at the time of radiographic disease progression, participants will be followed until they develop radiographic disease progression.

The study will be terminated early if less than 3 of the first 10 enrolled participants can complete 2 cycles of the adaptive abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate (the availability archival prostate tumor sample is preferred not required)
* Asymptomatic or minimally symptomatic (not requiring opioids for cancer related pain) metastatic castration resistant prostate cancer (CRPC) patients on abiraterone as standard of care and achieved at least 50% decline of their pre-treatment prostatic specific antigen (PSA)
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Adequate organ function
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections or major surgery within 28 days prior to study enrollment
* Prior surgical castration or concurrent use of gonadotropin-releasing hormone (GnRH) analogue (i.e. medical castration) with testosterone at screening <50 ng/dL.
* Ability to give written informed consent

Exclusion Criteria:

* Except GnRH analogue therapy, any other therapies for prostate cancer (excluding bisphosphonate and denosumab) must be discontinued 3 weeks before the first dose of study drugs.
* Prior treatments with Cyp 17 inhibitors like TAK-700/Orteronel, ketoconazole, radium 223 or docetaxel (up to 6 cycles of docetaxel given in the non CRPC setting is allowed). Prior treatment with Sipuleucel-T is allowed.
* Documented central nervous system (CNS) metastases or liver metastasis
* Treatment with any investigational compound within 30 days prior to the first dose of study drugs
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs, or previously diagnosed with another malignancy & have any evidence of residual disease. Potential participants with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Uncontrolled hypertension despite appropriate medical therapy (blood pressure of greater than 160 mmHg systolic and 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the Screening period). Note: May be rescreened after adjustments of antihypertensive medications
* Unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 [National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03], New York Heart Association (NYHA) Class III or IV heart failure
* Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C not contained with anti-viral therapy, life threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in investigator's opinion, potentially interfere with participation in this study.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of study drugs, including difficulty swallowing tables
* Delayed healing of wounds, ulcers, and/or bone fractures
* Inability to comply with protocol requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Prostatic Specific Antigen (PSA) Response Rate | End of cycle 2: 2 months per participant
  PSA response rate (defined as 50% decline of pre abiraterone PSA) at cycle 2. Rate in black participants, non-black participants, and participants overall.

SECONDARY OUTCOMES:
Median Radiographic Progression-Free Survival (rPFS) | Up to 36 months
  Radiographic progression defined by any of the following: 1.) Progression of measureable lesions per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over pretreatment baseline if no decrease during therapy) using the same imaging techniques as baseline, as well as an absolute increase of at least 0.5 cm. 2.) Progression on bone scan is defined as 2 or more new lesions on radionuclide bone scans. 3.) Unequivocal progression evidenced by appearance of 2 or more new measurable lesions at least 2 cm in short axis. Rate in black participants, non-black participants, and participants overall.
Median Time to Performance Status Deterioration | Up to 36 months
  Median Time to Eastern Cooperative Oncology Group (ECOG) Performance status in deterioration. 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work; 2- Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours; 3 - Capable of limited self-care, confined to bed or chair more than 50% of waking hours; 4 - Completely disabled; cannot carry on any self-care; totally confined to bed or chair. Rate in black participants, non-black participants, and participants overall.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Zhang J, Cunningham JJ, Brown JS, Gatenby RA. Integrating evolutionary dynamics into treatment of metastatic castrate-resistant prostate cancer. Nat Commun. 2017 Nov 28;8(1):1816. doi: 10.1038/s41467-017-01968-5. PMID 29180633